CLINICAL TRIAL: NCT06704958
Title: Augmented Momentary Personal Ecological Risk Evaluation
Acronym: AMPERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ian Bennett, Professor: Psychiatry & Behavioral Sciences, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00017404; P50MH129708-02 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Suicidal Ideation; Self Harm
Keywords: suicidal ideation; self harm
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Iterative intervention Development
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of AMPERE EMA prototype (Other): An EMA risk monitoring system using a smartphone EMA app to collect self-reported data from participating patients experiencing suicidal ideation.
  Interventions: Other: AMPERE EMA app

INTERVENTIONS:
Other: AMPERE EMA app — AMPERE EMA smartphone app using MyCap

SUMMARY:
The goal of this intervention study is to co-design and test an Ecological Momentary Assessment (EMA) prototype tool with young adults aged 16-30 experiencing suicidality to see if it is an acceptable and usable clinical tool for risk management.

The main study aims are:

* To co-design a prototype EMA suicide risk monitoring system with patients and health care provider input using Human Centered Design (HCD) methods.
* To test the developed EMA protype with providers and their young adult patients aged 16-30 experiencing suicidality to determine if the EMA prototype is an acceptable and usable clinical tool.

Young adult participants receiving care for active suicidal ideation will

* Download and use the EMA prototype for a total of two months.
* Complete 3 online surveys at 0, 1 and 2 months after enrolled in the study.

DETAILED DESCRIPTION:
Death by suicide is a leading cause of preventable mortality for young adults in the United States, yet the health care delivery system is poorly equipped to address this preventable issue. Ecological momentary assessment (EMA) allows patients to easily self-monitor and track symptoms using devices young adults already use (e.g., smartphones) in their natural environments, and can combine self-reported assessment with digital indicators of wellbeing via native smartphone sensors (e.g., daily step counts; number of device unlocks during the night, which may indicate sleep problems). EMA suicide risk detection systems show promise, but acceptability among patients at risk for suicide is unknown, and an actionable system for response to these signals by outpatient health care providers has not been developed.

The current project aims to design (Aim 1) and to examine the acceptability and feasibility of an EMA tool with young adults at risk of suicide in typical outpatient medical settings (Aim 2). Specifically, the goal of this intervention study is to see how EMA based signals of suicide risk can be used in primary health care to support management and care of young adults aged 16-30 experiencing suicidality. We will use human centered design (HCD) to co-develop and test an EMA protype with young adult patients and their health care providers to determine if acceptable and usable clinical tool. The goal of the project is to develop an EMA based prototype that improves management and care for young adults experiencing suicidality and has the potential to be used in other effective risk monitoring strategies to follow.

The specific aims of this proposed study are:

Aim 1: Co-design a prototype EMA suicide risk monitoring system with patients and health care providers through human centered design (HCD).

Aim 1.1 Iteratively co-design an EMA prototype with patient and providers; Aim 1.2 Develop training, and support materials for EMA clinical use. Aim 2: Conduct a feasibility and acceptability pilot of the EMA prototype to inform its revision and further development.

The pilot will consist of approximately 50 University of Washington Primary Care (UWPC) patients receiving care for active suicidal ideation in a UWPC clinical site. Following consent, the pilot participants will download the EMA prototype to their smart phone and use it for two months. During the two months, participants will use the EMA prototype to complete a weekly depression screener and brief daily surveys on mood, activity level, sleep, diet, substance use and social support. Patient participants will be asked to complete three online surveys, one right after they enroll, one at 1 month and one at 2 months following enrollment. The surveys will ask about demographic information (age, race, ethnicity, etc.), suicidal ideation, self-injury, substance use, social support and their experience using the EMA prototype.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (age 16-30 years)
* Receiving care at University of Washington Primary Care for suicidal ideation as determined by Electronic Health Record problem list or PHQ-9 suicide risk item >0 in previous year and/or recent (past year) history of suicide attempt and/or active suicidal ideation.
* Ability to consent to participate

Exclusion Criteria:

* Age <16 or >30,
* Non-English speaking
* No smart phone access
* Any clinical medical/psychiatric condition, severity of that condition, or life situation that would compromise safe and voluntary study participation.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Scale (AIM) | 2 month post-initiation of AMPERE EMA use
  This is a four-item measure of intervention acceptability, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. Total mean scores range from 1 - 5, with higher scores indicating higher acceptability. Participants will complete this measure after 4 weeks of using the mobile mental health app to which they are randomized.
System Usability Scale (SUS) | 2 month post-initiation of AMPERE EMA use
  This is a 10 item measure of system usability with 5 response options. SUS score can range from 0 to 100 with a higher score indicating high usability.
Client Satisfaction Questionnaire (CSQ) | 2 month post-initiation of AMPERE EMA use
  This is a 3 item measure to assess consumer satisfaction with health and human services

SECONDARY OUTCOMES:
Suicide Related Coping Scale (SRCS) | 0, 1, 2 month post-initiation of AMPERE EMA use
  Suicide-Related Coping Scale (SRCS) measures how well a person manages suicidal thoughts through the use of internal and external coping strategies. A 17-item tool with two score factors, internal and external coping strategies.
Helping Alliance Questionnaire (Haq-II) | 1, 2 month post-initiation of AMPERE EMA use
  The Helping Alliance Questionnaire is a 11-item patient self-report measure which assesses the extent to which the patient experiences the therapist and the therapy as helpful. It contains two types of helping alliance: Type I -- Perceived Helpfulness -- defined as the patient's experience of the therapist as providing or being capable of providing the help that is needed; and Type II -- Collaboration or Bonding -- defined as the patient's experience of treatment as a process of working together with the therapist toward the goals of treatment. The HAQ contains 11 items rated on a 4-point scale (completely disagree, disagree, agree, and completely agree).

OTHER OUTCOMES:
PhenX Social Determinants of Health Core | 0 month post-initiation of AMPERE EMA use
  The PhenX Social Determinants of Health (SDOH) Collection is a toolset to help measure individual as well as structural factors that shape behaviors and health outcomes. The Core Collection is designed to create common data elements for measuring key variables across studies or clinical trials. It includes elements such as: Race and Ethnicity, Age, Gender Identity, Annual Family Income, English Proficiency, Occupational Prestige and Access to Health Services.
Patient Health Questionnaire (PHQ-9) | 0 month post-initiation of AMPERE EMA use
  The Patient Health Questionnaire (PHQ-9) consists of 9 depression items and one disability item. Each item is associated with a DSM symptom of depression, which the participant rates whether or not they have experienced the symptom over the last two weeks, with severity rating of 0-3. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time, with a total sum score ranging from 0 - 27. Higher scores indicate higher depression symptom severity.
Generalized Anxiety Disorder (7-Item) Scale (GAD-7) | 0 month post-initiation of AMPERE EMA use
  The Generalized Anxiety Disorder Scale (GAD-7) is a 7- item screener for generalized anxiety. It consists of items related to generalized anxiety disorder. Participants rate on a scale of 0-3 how much they have experienced in the last two weeks to crease a total sum score ranging from 0 - 21. The scale is a valid screener for generalized anxiety symptoms. Higher scores indicate higher anxiety symptom severity.
WHO ASSIST V3.0 | 0 month post-initiation of AMPERE EMA use
  World Health Organization (WHO) Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) is a questionnaire that screens for all levels of problem or risky substance use in adults. The ASSIST consists of eight questions covering tobacco, alcohol, cannabis, cocaine, amphetamine-type stimulants (including ecstasy) inhalants, sedatives, hallucinogens, opioids and 'other drugs'. A risk score is provided for each substance, and scores are grouped into 'low risk', 'moderate risk' or 'high risk'. The risk score determines the level of intervention recommended (brief intervention or brief intervention plus referral to specialist treatment).
EuroQol 5 Dimension Youth (EQ-5D-Y) | 0 month post-initiation of AMPERE EMA use
  EQ-5D is a standardized measure of health-related quality of life. The EQ-5D-Y was adapted from the EQ-5D to assess health-related quality of life (HRQOL) for use in children and adolescents. The standard adult EQ-5D consists of a descriptive system that comprises five items referring to the domains mobility, self-care, usual activities, pain/discomfort and anxiety/depression scored as presenting no problems, moderate problems or severe problems.
Columbia Suicide Severity Rating Scale Screener (C-SSRS) | 0, 1, 2 month post-initiation of AMPERE EMA use
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a suicide risk assessment tool that supports suicide risk assessment through a series of simple, plain-language questions. The answers help users identify whether someone is at risk for suicide, assess the severity and immediacy of that risk, and gauge the level of support that the person needs. This scale allows scores from 0-6.
Harkavy Anais (HASS) Ideation | 0, 1, 2 month post-initiation of AMPERE EMA use
  The Harkavy Asnis Suicide Survey (HASS), a self-report instrument designed to gather detailed information regarding demographics, past suicidal behavior (SB) in patients as well as their family and associates, and current SB. The HASS may be helpful in assessing the whole spectrum of SB (from ideation to attempts) in psychiatric patients of all diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Bennett, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided